CLINICAL TRIAL: NCT04850105
Title: A Prospective, Non-interventional, Long-term, Multinational Cohort Safety Study of Patients With Hereditary Transthyretin Amyloidosis With Polyneuropathy (hATTR-PN)
Brief Title: A Non-interventional Cohort Safety Study of Patients With hATTR-PN
Status: Recruiting | Type: Observational
Sponsor: Akcea Therapeutics (Industry)
Collaborators: United BioSource, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: TEG4001; EUPAS37728 (Other: EU PAS)
Record Dates: First submitted 2021-04-06; First posted 2021-04-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Transthyretin Amyloidosis With Polyneuropthy
Keywords: Hereditary Transthyretin Amyloidosis; hATTR-PN; hATTR; Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TEGSEDI-exposed cohort: This cohort consist of patients diagnosed with hATTR-PN who are receiving any dose of commercial TEGSEDI and who have provided written informed consent to be included into the study.
  Interventions: Other: Data Collection
- TEGSEDI-unexposed cohort: This cohort which will consist of patients diagnosed with hATTR-PN who have not taken any dose of TEGSEDI within 25 weeks prior to enrollment and are eligible for TEGSEDI treatment per applicable product label and who have provided written informed consent to be included into the study.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Data on each patient will be collected at study enrollment and at each follow-up visit.
  No mandatory visits, tests, or assessments are required for this study. All visits will be scheduled and conducted according to the clinical site's normal clinical practice.

SUMMARY:
This is a prospective, non-interventional, Long-term, multinational cohort safety study of patients with Hereditary Transthyretin Amyloidosis with Polyneuropathy (hATTR-PN). The overarching goal of this study is to further characterize the long-term safety of TEGSEDI (inotersen) in patients with hATTR-PN under real-world conditions.

DETAILED DESCRIPTION:
Study Rationale:

hATTR-PN is an inherited, progressive, fatal disease caused by misfolded transthyretin (TTR) proteins that accumulate as amyloid fibrils predominantly in the peripheral nerves, heart, gastrointestinal tract, and other organs. hATTR-PN is a rare disease and there are no large epidemiological studies that reliably provide an indication of its prevalence. The worldwide distribution is unequal, with higher rates in Portugal, Japan, Northern Sweden, and the US. Current estimates suggest there may be 10,000 afflicted patients worldwide.

TEGSEDI (inotersen) is an antisense oligonucleotide inhibitor of human TTR protein synthesis. In Europe and Canada, TEGSEDI is indicated for the treatment of Stage 1 or Stage 2 polyneuropathy in adult patients with hereditary transthyretin amyloidosis (hATTR). In the US, TEGSEDI is indicated for treatment of the polyneuropathy of hereditary TTR-mediated amyloidosis in adults. Efficacy has been demonstrated in patients with hATTR-PN, as reflected by a slowing or reversal of disease progression.

Research Question:

The overarching goal of this study is to further characterize the long-term safety of TEGSEDI in patients with hATTR-PN under real-world conditions.

Population:

Patients in Europe, US, and Canada will be enrolled from centers that manage patients with hATTR-PN. Physicians participating in the study will be instructed to invite all patients who meet study eligibility criteria to enroll until the enrollment period is closed.

ELIGIBILITY:
Inclusion Criteria:

1. Either:

   1. TEGSEDI Exposed Cohort: Patients diagnosed with hATTR-PN who have taken any dose of TEGSEDI within 25 weeks prior to enrollment
   2. TEGSEDI Unexposed Cohort: Patients diagnosed with hATTR-PN who have not taken any dose of TEGSEDI within 25 weeks prior to enrollment and are eligible for TEGSEDI treatment per applicable product label. Patients may take other drugs to treat hATTR-PN.
2. Clinically managed in Canada, Europe, or the US
3. Have provided appropriate written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The TEGSEDI-exposed cohort will consist of patients diagnosed with hATTR-PN who are receiving TEGSEDI. Data from the TEGSEDI-exposed cohort will be compared to data collected prospectively from a TEGSEDI-unexposed cohort which will consist of patients diagnosed with hATTR-PN who have not taken any dose of TEGSEDI within 25 weeks prior to enrollment and are eligible for TEGSEDI treatment per applicable product label.
  Patients in Europe, US, and Canada will be enrolled from centers that manage patients with hATTR-PN.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2036-03-31 (Estimated); Study Completion 2036-03-31 (Estimated)

PRIMARY OUTCOMES:
Further characterization of the long-term safety of TEGSEDI in patients with hATTR-PN under real-world conditions. | 10 years
  * Determination of the incidence rate of thrombocytopenia in patients with hATTR-PN treated with TEGSEDI (TEGSEDI-exposed cohort)
  * Comparison of the relative rates of thrombocytopenia in hATTR-PN patients treated with TEGSEDI (TEGSEDI exposed) to hATTR-PN patients unexposed to TEGSEDI (TEGSEDI- unexposed)

SECONDARY OUTCOMES:
Description of the incidence rate of the Adverse Events of Special Interest (AESI) in the TEGSEDI-exposed and TEGSEDI-unexposed patients. | 10 years
  To describe the incidence rate of the following Adverse Events of Special Interest (AESI):
  * severe thrombocytopenia (platelet counts <25 x 109/L and separately, <50 x 109/L)
  * serious and non-serious bleeding events
  * glomerulonephritis
  * hepatotoxicity/serious hepatobiliary events
  * composite of stroke and/or cervicocephalic arterial dissection
  * central nervous system (CNS) vasculitis
  * ocular toxicity due to vitamin A deficiency
Description of the time to onset of Adverse Events of Special Interest (AESI) in the TEGSEDI-exposed and TEGSEDI-unexposed patients. | 10 years
  To describe the time to onset of the following Adverse Events of Special Interest (AESI):
  * severe thrombocytopenia
  * serious and non-serious bleeding events
  * glomerulonephritis
  * hepatotoxicity/serious hepatobiliary events
  * composite of stroke and/or cervicocephalic arterial dissection
  * central nervous system (CNS) vasculitis
  * ocular toxicity due to vitamin A deficiency

CONTACTS AND LOCATIONS:
Locations (24):
- Study Centre, Sofia, Bulgaria
- Study Centre, Égkomi, Nicosia, Cyprus
- France (3):
  - Study Center, Lille, Cedex
  - Study Center, Nice, Romaine
  - Study Centre, Nantes
- Study Center, Heidelberg, Germany
- Greece (2):
  - Study Center, Athens
  - Study Center, Heraklion
- Italy (8):
  - Study Centre, Roma, Rome
  - Study Center, Bologna
  - Study Center, Genova
  - Study Center, Messina
  - Study Center, Milan
  - Study Center, Napoli
  - Study Center, Pavia
  - Study Center, Roma
- Study Center, Lisbon, Portugal
- Spain (7):
  - Study Center, Huelva, Andalusia
  - Study Centre, Oviedo, Avenida de Roma
  - Study Center, Palma de Mallorca, Balearic Islands
  - Study Centre, Villarreal, Barcelona
  - Study Centre, Barcelona, Catalonia
  - Study Centre, Madrid, Madrid
  - Study Center, Madrid

IPD SHARING:
Plan to Share IPD: No